CLINICAL TRIAL: NCT05401279
Title: Bladder Sparing Treatment of Tislelizumab Combined With Gemcitabine and Cisplatin for Patients With PD-L1 Positive Muscle Invasive Bladder Cancer (T2-3N0M0): a Phase II Prospective Study
Brief Title: Bladder Sparing Treatment of Tislelizumab, Gemcitabine and Cisplatin for Patients With PD-L1 Positive Muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TICIG
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Urothelial Carcinoma Bladder; PD-1 Inhibitor
MeSH Terms: interventions — tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine, Cisplatin and Tislelizumab (Experimental): Patients will receive transurethral resection or partial cystectomy to remove all visible tumors with no residual disease left. 2-4 weeks after the surgery, patients will receive 8 cycles of tislelizumab combined with 4-6 cycles of gemcitabine and cisplatin.
  Interventions: Drug: Tislelizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg will be administered on Day 1 of each 21 day cycle for 8 21-day cycles.
Drug: Gemcitabine — Gemcitabine 1000mg/m^2 will be administered on Days 1 and 8 for four to six 21-day cycles.
Drug: Cisplatin — Cisplatin 70mg^m2 will be administered on Day 1 for four to six 21-day cycles.

SUMMARY:
This is a phase II open label single-arm prospective study aiming to investigate the efficacy of PD-1 inhibitor Tislelizumab combined with conventional gemcitabine and cisplatin as bladder sparing treatment for patients with PD-L1 positive muscle invasive bladder carcinoma (T2-3N0M0).

DETAILED DESCRIPTION:
The study will enroll 20 patients with adequate organ function and performance status who either wish to attempt bladder preserving therapy or are ineligible for radical cystectomy. The bladder samples must be available and assessed as positive for PD-L1 expression . Patients will receive transurethral resection or partial cystectomy to remove all visible tumors with no residual disease left. After the surgery, patients will receive 8 cycles of tislelizumab combined with 4-6 cycles of gemcitabine and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed muscle-invasive urothelial cancer of the bladder within 60 days of study enrollment. Variant histology and cis are not allowed. Patients must be willing to provide a TURBT specimen during screening and prior to enrollment if adequate specimen (FFPE tissue block or 20 unstained slides) from initial TURBT documenting muscle-invasive urothelial bladder cancer is not available. The specimen must be assessed as PD-L1 positive by two pathologists using SP263 kit.
2. Clinical stage T2-T3, N0, M0 urothelial bladder cancer.
3. Deemed to not be a candidate for radical cystectomy by attending urologic oncologist or refuse radical cystectomy.
4. Willing to receive maximal transurethral resection or partial cystectomy to remove all bladder tumors
5. Be willing and able to provide written informed consent/assent for the trial.
6. Have a performance status of 0 or 2 on the Eastern Cooperative Oncology Group Performance Scale.
7. Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days of protocol enrollment.

   * Absolute neutrophil count >= 1,500 /mcL;
   * Platelets >= 100,000 /mcL;
   * Hemoglobin >= 9.0 g/dL;
   * Serum creatinine <=1.5 x upper limit of normal (ULN) or calculated creatinine clearance >= 30 mL/min as calculated by Cockcrof-Gault formulae or by 24 hour urine collection;
   * Serum total bilirubin <=1.5 x ULN or direct bilirubin <= ULN for subjects with total -bilirubin levels > 1.5 x ULN;
   * Aspartate aminotransferase and alanine aminotransferase <= 1.5 x ULN;
   * Albumin >= 2.5 mg/dL;
   * International normalized ratio or prothrombin time (PT) <= 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial prothrombin time (PTT) is within therapeutic range of intended use of anticoagulants;
   * Activated Partial Thromboplastin Time (aPTT) <= 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Has received prior radiation therapy or systemic chemotherapy for urothelial bladder cancer including neoadjuvant chemotherapy. Prior intravesical chemotherapy or intravesical immunotherapy is permissible, however, no prior intravesical therapy is permitted within 4 weeks of study enrollment; adjuvant therapy is not permitted.
2. Has received prior pelvic radiation therapy.
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
5. Has a known history of active TB (Bacillus Tuberculosis).
6. Hypersensitivity to tislelizumab or any of its excipients.
7. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Any prior history of invasive malignancy within the past 5 years except non-melanoma skin cancer, carcinoma in-situ, localized prostate cancer without biochemical recurrence following definitive treatment.
10. Has other active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. History of Guillain-Barre Syndrome or Stevens-Johnson Syndrome
12. Has known history of, or any evidence of active, non-infectious pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
20. Has received a live vaccine within 30 days of planned start of study therapy. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Two-year bladder-intact disease-free survival rate | 2 years
  Bladder-intact disease-free survival is defined as time from initiation of protocol therapy until the development of muscle-invasive bladder cancer recurrence, regional pelvic recurrence, distant metastases, bladder cancer-related death, or cystectomy.

SECONDARY OUTCOMES:
Adverse Events | 2 years
  The adverse events are evaluated per Common Terminology Criteria for Adverse Events (CTCAE) 5.
Overall survival | up to 5 years
  Defined as time to death from beginning of protocol therapy
Metastasis-free survival | up to 5 years
  Defined as time to the development of radiographic distant metastases from beginning of protocol therapy.
Disease-free survival | up to 5 years
  Defined as time to recurrence, metastasis or death from beginning of protocol therapy.
Disease specific survival | up to 5 years
  Defined as time to death because of bladder cancer from beginning of protocol therapy

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xue, PhD, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No